CLINICAL TRIAL: NCT00310479
Title: Clinico-pathologic Correlative Study of 3T Magnetic Resonance Spectroscopy in the Localization of Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GU-6-0062 / 22281
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: Magnetic Resonance Imaging; prostate cancer imaging; 3T MRS; functional imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Magnetic Resonance Spectroscopy (3Tesla)

SUMMARY:
We seek to develop an advanced imaging approach to identifying and localizing prostate cancer. We believe that high field MRI (magnetic resonance imaging) has the potential to do this and we will endeavor to prove this by having patients with prostate cancer pre-operatively undergo a technique called magnetic resonance spectroscopy. After surgery, the microscopic locations of cancer will be compared with the pre-operative images to assess how well the imaging technique succeeds.

DETAILED DESCRIPTION:
The proposed research is enormously relevant to the clinical understanding of early prostate cancer. We propose to test to see whether characteristic patterns of invivo 3T MRSI associated metabolites can be identified in correlation with clinically active tumor reserved on histopathologic analysis of resected specimens. We also plan to demonstrate that 3T MR spectra of prostate cancer will allow for more detailed metabolic assessment with higher sensitivity, specificity and accuracy and publish results established from MR spectra using 1.5T MR units. Functional imaging (eg. molecular imaging such as this) is felt to be the clinical wave of the future for cancer imaging, and if successful, will assume a very major role in the detection, assessment, treatment planning and delivery of drugs, radiation, heat and novel therapeutics in the fight against prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified prostate cancer
* Patient has opted for surgery
* Low risk prostate cancer PSA <1 0, Gleason < 7, Stage < T2b
* No contraindication to MR scanning
* No prior history of malignancy
* Fit for surgery

Exclusion Criteria:

* Nonbiopsied lesion
* Intermediate or high risk prostate cancer
* Unfit for surgery
* Contraindication to MR scanning (i.e. pacemaker, aneurysm clips, claustrophobia)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
characteristic metabolic pattern of prostate cancer at 3Tesla

SECONDARY OUTCOMES:
specificity, accuracy, NPV
PPV of MRS in the detection of prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Parliament, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada